CLINICAL TRIAL: NCT05792813
Title: Xiyuan Hospital of China Academy of Chinese Medical Sciences
Brief Title: Efficacy and Safety of Linggui Yangyuan Paste in Patients With Male Infertility
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other); Shandong University of Traditional Chinese Medicine (Other); Chengdu Fifth People's Hospital (Other); Affiliated Hospital of Nanjing University of Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Xiyuannanke
Record Dates: First submitted 2023-03-08; First posted 2023-03-31 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-03

CONDITIONS: Male Infertility; Asthenozoospermia; Oligoasthenozoospermia
MeSH Terms: conditions — Infertility, Male; Asthenozoospermia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): LGYY+ WZYZ mimetic
  Interventions: Drug: LGYY; Drug: WZYZ mimetic
- Control group (Active Comparator): WZYZ + LGYY mimetic
  Interventions: Drug: LGYY mimetic; Drug: WZYZ

INTERVENTIONS:
Drug: LGYY — LGYY = Linggui Yangyuan paste
  Arms: Experimental group
Drug: LGYY mimetic — LGYY = Linggui Yangyuan paste
  Arms: Control group
Drug: WZYZ — WZYZ= Wuzi Yanzong oral solution
  Arms: Control group
Drug: WZYZ mimetic — WZYZ= Wuzi Yanzong oral solution
  Arms: Experimental group

SUMMARY:
Male infertility affects millions of males worldwide and is rising in prevalence due to social and environmental conditions. Asthenozoospermia (AZS) and oligoasthenozoospermia (OA) are the major causes of male infertility. The diagnosis of male infertility has a negative effect on men's physical and psychological status, poses a threat to their social relationships, lowers self-esteem, and disrupts family harmony. At present, the treatment of ASZ and OA are all mostly empirical, including antioxidants, endocrine therapy, and anti-infection. However, there are still limitations due to inefficiencies. Linggui Yangyuan paste (LGYY), a traditional Chinese compound herbal past, had been used to treat ASZ and OA for several years at the Xiyuan Hospital of China Academy of Chinese Medical Sciences. The investigators designed this program to study the efficacy and safety of LGYY for the treatment of patients with male infertility (AZS and OA).

ELIGIBILITY:
Inclusion Criteria:

* The participants must meet all following criteria at the time of randomization to be eligible for recruitment :

  1. Study participants met the diagnostic criteria for male infertility 1)inability to have a child after at least 1 year of marriage with regular sexual life and without using any preventive methods 2)normal fertile female partner
  2. Study participants met the diagnostic criteria for AZS or OA

For AZS:

1. sperm concentration ≥15 × 106/ mL
2. PR <32%

For OA:

1. sperm concentration <15 × 106/ mL
2. PR <32% (3) Study participants met the TCM diagnosis criteria for kidney deficiency and blood stasis (4) Men aged 22 to 45 years (5) The participants signed informed consent forms

Exclusion Criteria:

* The trial exclusion criteria included any of the following:

  1. infertility is caused by the inability to complete sexual intercourse, including but not limited to erectile dysfunction or ejaculatory disorders
  2. with infertility caused by organic lesions of the reproductive system
  3. with reproductive system infection, such as chlamydia trachomatis or mycoplasma infection
  4. with palpable varicocele
  5. with abnormal and clinical significance of sex hormone (FSH, LH, T)
  6. complicated with liver and kidney dysfunction, severe basic diseases such as diabetes, cardiovascular and cerebrovascular diseases, mental diseases, malignant tumors, or serious organic diseases
  7. with a history of allergy to any medicine or ingredients used in this study
  8. receive other relevant treatment for the disease 2 weeks before treatment

Ages: 22 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 162 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Total progressive motile sperm count (TPMSC) from baseline to post-treatment | Baseline, 12 weeks
  TPMSC change from baseline to post-treatment

SECONDARY OUTCOMES:
The total sperm count change from baseline to post-treatment | Baseline, 4, 8, 12 weeks
  the total sperm count change from baseline to post-treatment
semen volume change from baseline to post-treatment | Baseline, 4, 8, 12 weeks
  1) semen volume
sperm density change from baseline to post-treatment | Baseline, 4, 8, 12 weeks
  2) sperm density
PR rate change from baseline to post-treatment | Baseline, 4, 8, 12 weeks
  3) Semen parameter PR rate
PR+NP rate change from baseline to post-treatment | Baseline, 4, 8, 12 weeks
  4) PR+NP rate
Chinese Medicine Symptoms Score (CMSS) change from baseline to post-treatment | Baseline, 4, 8, 12 weeks of treatment and 12 weeks of follow-up (24 week)
  Scores range from 0 to 33 with higher scores indicating greater burden of symptoms.
spouse pregnancy rate | Baseline, 12 weeks of treatment and 12 weeks of follow-up (24 week)
  difference in the number of pregnancies
time to pregnancy | Baseline, 12 weeks of treatment and 12 weeks of follow-up (24 week)
  The time required for pregnancy in this study

IPD SHARING:
Plan to Share IPD: Undecided